CLINICAL TRIAL: NCT02057731
Title: Characterizing Expression of Glycogen Storage Disease in Heterozygous Carriers
Brief Title: Study of Glycogen Storage Disease Expression in Carriers
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201300688
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-12

CONDITIONS: Glycogen Storage Disease
MeSH Terms: conditions — Glycogen Storage Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Ia carriers: Carriers of GSD type Ia will have their blood and urine tested to measure markers of GSD. Their saliva will be tested to determine their specific mutation. A questionnaire will also be filled out.
  Interventions: Genetic: Glycogen Storage Disease markers
- Ib carriers: Carriers of GSD type Ib will have their blood and urine tested to measure markers of GSD. Their saliva will be tested to determine their specific mutation. A questionnaire will also be filled out.
  Interventions: Genetic: Glycogen Storage Disease markers
- III carriers: Carriers of GSD type III will have their blood and urine tested to measure markers of GSD. Their saliva will be tested to determine their specific mutation. A questionnaire will also be filled out.
  Interventions: Genetic: Glycogen Storage Disease markers
- 0, VI, IX carriers: Carriers of GSD types 0, VI, and IX will have their blood and urine tested to measure markers of GSD. Their saliva will be tested to determine their specific mutation. A questionnaire will also be filled out.
  Interventions: Genetic: Glycogen Storage Disease markers
- Noncarriers: Noncarriers of any type of GSD will have their blood and urine tested to measure markers of GSD. Their saliva will be tested to ensure their noncarrier status. A questionnaire will also be filled out.
  Interventions: Genetic: Glycogen Storage Disease markers

INTERVENTIONS:
Genetic: Glycogen Storage Disease markers — Blood and urine tests will be performed on all groups to measure markers of GSD. A saliva DNA test will be used to determine the specific mutation the carrier has or to ensure noncarrier status. A questionnaire will also be filled out.

SUMMARY:
The purpose of the study is to determine whether carrier status for any type of glycogen storage disease (GSD) predisposes the carrier to GSD markers, like high cholesterol, by testing blood, urine, and saliva samples.

DETAILED DESCRIPTION:
Subjects will be asked to contribute about a teaspoon of blood, 1 oz of urine, and 2 tablespoons of saliva samples in the morning before they have had anything to eat. The blood and urine samples will be tested for the markers of GSD, while the saliva sample will be used for genetic testing. Subjects' height and weight will also be measured.

Subjects will also be asked to fill out a questionnaire about symptoms common to full GSD expression that they may have experienced, as well as if they are currently on any medication to control their cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* parents and other family members of patients undergoing treatment for GSD at the University of Florida

Exclusion Criteria:

* pregnant females

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parents and other family members of patients currently undergoing treatment for GSD at the University of Florida
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2014-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Cholesterol level blood test | 1 day
  Blood test will be performed on all groups to measure markers of glycogen storage disease.

SECONDARY OUTCOMES:
Comprehensive metabolic panel blood test | 1 day
  Blood test will be performed on all groups to measure markers of glycogen storage disease.
Lipid panel blood test | 1 day
  Blood test will be performed on all groups to measure markers of glycogen storage disease.
Uric acid level blood test | 1 day
  Blood test will be performed on all groups to measure markers of glycogen storage disease.
Creatine kinase (CK) level blood test | 1 day
  Blood test will be performed on all groups to measure markers of glycogen storage disease.
C-reactive protein (CRP) level blood test | 1 day
  Blood test will be performed on all groups to measure markers of glycogen storage disease.
Calcium level urine test | 1 day
  Urine test will be performed on all groups to measure markers of glycogen storage disease.
Citrate level urine test | 1 day
  Urine test will be performed on all groups to measure markers of glycogen storage disease.
Creatinine level urine test | 1 day
  Urine test will be performed on all groups to measure markers of glycogen storage disease.
Microalbumin level urine test | 1 day
  Urine test will be performed on all groups to measure markers of glycogen storage disease.
Oxalate level urine test | 1 day
  Urine test will be performed on all groups to measure markers of glycogen storage disease.
Uric acid level urine test | 1 day
  Urine test will be performed on all groups to measure markers of glycogen storage disease.
Prealbumin blood test | 1 day
  Blood test will be performed on all groups to measure markers of glycogen storage disease.
Hemoglobin A1C blood test | 1 day
  Blood test will be performed on all groups to measure markers of glycogen storage disease.

CONTACTS AND LOCATIONS:
Overall Officials: David A Weinstein, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Weinstein DA, Correia CE, Conlon T, Specht A, Verstegen J, Onclin-Verstegen K, Campbell-Thompson M, Dhaliwal G, Mirian L, Cossette H, Falk DJ, Germain S, Clement N, Porvasnik S, Fiske L, Struck M, Ramirez HE, Jordan J, Andrutis K, Chou JY, Byrne BJ, Mah CS. Adeno-associated virus-mediated correction of a canine model of glycogen storage disease type Ia. Hum Gene Ther. 2010 Jul;21(7):903-10. doi: 10.1089/hum.2009.157. PMID 20163245